CLINICAL TRIAL: NCT01964833
Title: Combination of Photodynamic Therapy and Periodontal Treatment in Patients With Type 2 Diabetes Mellitus: Randomized, Double-blind Clinical Trial
Brief Title: PDT and Periodontal Treatment in DMT2 Patients
Acronym: PDTDMT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cristiane Miranda Franca, Professor of the Post Graduation Program of Biophotonics applied to Health Sciences, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 375.454; 375.454 (Other: University Nove de Julho Ethics Comittee)
Record Dates: First submitted 2013-10-10; First posted 2013-10-17 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Periodontitis; Diabetes Mellitus Type 2
Keywords: clinical trial; DMT2; periodontitis; PDT
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2 | interventions — Periodontal Index; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Periodontal treatment (Sham Comparator): Conventional periodontal treatment with hygiene orientation, calculus removal and root scaling and planing. Sham PDT.
  Interventions: Procedure: Periodontal treatment
- Periodontal Treatment and PDT (Experimental): Conventional periodontal treatment with hygiene orientation, calculus removal, root scaling and planing. Active PDT with diode laser and methylene blue photosensitizer
  Interventions: Procedure: Periodontal treatment and PDT

INTERVENTIONS:
Procedure: Periodontal treatment — Periodontal treatment will consist of oral hygiene instructions, with the monitored orientation of brushing technique and recommendation of the daily use of dental floss. Calculus deposits will also be removed using ultrasound equipment with the appropriate tips for periodontics as well as scaling and planing with dental instruments, as recommended by the AAP (2001). Treatment will be carried out in two to four one-hour sessions.
  Patient will receive sham PDT.
  Arms: Periodontal treatment
Procedure: Periodontal treatment and PDT — Patients will receive periodontal treatment as previously described and PDT. PDT will be administered at the end of the periodontal treatment session at sites with pocket depths equal to or greater than 4 mm. A diode laser will be used at the 660 nm wavelength, P= 100 mW, 9 J/point, D = 22 J/cm2 (per point). The photosensitizer (BlueMet 0.005 % DMC)will be deposited at the fundus of the periodontal pocket using a syringe. The laser will be applied to the mucosa over the oral epithelium that lines the periodontal pocket using an optical fiber.
  Arms: Periodontal Treatment and PDT

SUMMARY:
The relationship between diabetes mellitus (DM) and periodontal disease is bidirectional. DM is a predisposing and modifying factor of periodontitis, which, in turn, worsens glycemic control and increases proteins found in the acute phase of inflammation. The gold standard for the treatment of periodontal disease is oral hygiene orientation, scaling and planing. Moreover, systemic antibiotic therapy may be employed in some cases. In an effort to minimize the prescription of antibiotics, photodynamic therapy (PDT) has been studied as an antimicrobial technique and has demonstrated promising results. The aim of the proposed study is to determine whether PDT as a complement to periodontal therapy (PT) is helpful in the metabolic control of individuals with type 2 diabetes and the reduction of acute phase inflammatory markers. The patients will be randomized using a proper software program into two groups: 1) PT + placebo PDT or 2) PT + active PDT. All patients will first be examined by a specialist, followed by PT performed by two other healthcare professionals. At the end of each session, PDT (active or sham) will be administered by a fourth healthcare professional. The following will be the PDT parameters: diode laser (660 nm); power output = 110 mW; exposure time = 90 seconds per point (9 J/point); and energy density = 22 J/cm2. The photosensitizer will be methylene blue (50 µg/mL). The patients will be re-evaluated 15, 30, 90 and 180 days after treatment. Serological exams with complete blood count, fasting glucose, glycated hemoglobin and crevicular fluid exams to screen for tumor necrosis factor alpha, interleukin 1, interleukin 6, osteocalcin, osteoprotegerin/RANKL will be performed at each evaluation. At baseline and 180 day periapical radiographs will be performed to evaluate the alveolar bone crest level. The data will be statistically evaluated using the most appropriate tests.

DETAILED DESCRIPTION:
Randomization of the patients to the different groups will be performed with the appropriate software program. Only the lead researcher will have access to the randomization list. Allocation to the two groups will be carried out in blocks of four.

The patients will be sent to Operator A for the periodontal exam. Without knowledge of the results of this exam, the patients will be treated by Operators B and C for periodontal treatment, which will involve oral hygiene instructions as well as supra-gingival and sub-gingival scaling and planing in up to four sessions. At the end of each session, the patients will be sent to Operator D, who will administer either placebo or active PDT based on the content of the sealed envelope. Thus, both the patients and operator in charge of the periodontal exams will be blinded to the PDT protocol (double-blind study).

Fasting blood sugar and glycated hemoglobin exams will be performed at baseline as well as 15, 30, 90 and 180 days after the completion of treatment. All exams will be carried out at the same laboratory affiliated with the university.

The clinical periodontal exams will be performed by a single examiner specialized in periodontics, who will evaluate six regions of each tooth with a 15-mm probe (North Carolina model, Hu-Friedy, Chicago, IL, USA). The following aspects will be recorded: plaque index, bleeding upon probing, probing depth, gingival recession and attachment loss (Armitage, 2004). Evaluations will be carried out performed at baseline (prior to initial treatment) as well as 15, 30, 90 and 180 days after the completion of treatment.

Patients will receive periodontal treatment and photodynamic therapy (active or sham depending on the allocation).

Crevicular fluid will be collected from the previously defined sites with a probing depth equal to or greater than 4 mm that will receive treatment. Collection will be performed with relative isolation using cotton rolls following the removal of supra-gingival plaque with periodontal curettes and air drying for five seconds. Absorbent paper strips (PerioPaper, ProFlow Inc., Amityville, NY, USA) will be individually inserted into each site for 30 seconds (Rudin et al., 1970). The collections will be performed by a single researcher. The volume of crevicular fluid samples will be measured using the Periotron 8000 micro-moisture meter (Oraflow Inc., NY, USA). The samples will then be placed in duly identified sterile plastic microtubes, temporarily stored in dry ice and subsequently stored in a freezer at -80 ºC

ELIGIBILITY:
Inclusion Criteria:

1. Compensated type 2 diabetes mellitus or with adequate control based on the criteria of the Brazilian Society of Diabetes (SBD, 2012);
2. Chronic periodontitis (AAP, 2001);
3. Presence of at least 15 teeth and at least four teeth with bleeding upon probing and probing depth greater than 4 mm;
4. Aged 18 years or older;
5. Under follow up with an endocrinologist.

Exclusion Criteria:

1. Uncompensated diabetes, based on SBD criteria;
2. Smoking habit in 12 months prior to treatment;
3. Anemia;
4. Active cancer;
5. Current pregnancy;
6. History of antibiotic therapy in previous six months;
7. History of anti-inflammatory therapy in previous three months;
8. Clotting disorder (use of anti-coagulant, presence of liver disease, thrombocytopenia and immunosuppression);
9. Currently undergoing orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in the clinical attachment level at 180 days. | 180 days
  Clinical attachment level is the depth measured from the CEJ (cement-enamel junction) to the bottom of the gingival sulcus. It indicates the amount of attachment that has been lost.

SECONDARY OUTCOMES:
Changes in the fasting blood and glycated hemoglobin (HBA1C) | Baseline, 15, 30, 90 and 180 days
  These tests reflects the glycemic control at the moment of the dental exam and the average blood sugar level for the past two to three months.
Cytokines in the crevicular fluid | Baseline, 15, 30, 90 and 180 days
  The crevicular fluid will be collected and investigated for the presence of IL-1, IL-6, TNF-alfa, osteocalcin, osteoprotegerin/RANKL in the crevicular fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane M Franca, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Evangelista EE, Franca CM, Veni P, de Oliveira Silva T, Goncalves RM, de Carvalho VF, Deana AM, Fernandes KP, Mesquita-Ferrari RA, Camacho CP, Bussadori SK, Alvarenga LH, Prates RA. Antimicrobial photodynamic therapy combined with periodontal treatment for metabolic control in patients with type 2 diabetes mellitus: study protocol for a randomized controlled trial. Trials. 2015 May 27;16:229. doi: 10.1186/s13063-015-0757-3. PMID 26013003